CLINICAL TRIAL: NCT00957307
Title: Breast CT as a Diagnostic Tool
Brief Title: Breast Computed Tomography (CT) as a Diagnostic Tool
Status: Completed | Type: Observational
Sponsor: Emory University (Other)
Responsible Party: Principal Investigator, Ioannis Sechopoulos, Ph.D., Assistant Professor of Radiology and Imaging Sciences, Emory University
Other Study IDs: IRB00014006
Record Dates: First submitted 2009-08-11; First posted 2009-08-12 (Estimated); Last update posted 2015-07-23 (Estimated); Status verified 2015-07

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Lay Summary

The American Cancer Society has recommended that all women over the age of 40 have an annual mammogram for many years. This recommendation has been associated with a substantial decrease in breast cancer deaths. When something suspicious is seen in one of these mammograms, the woman is called back to the clinic for more imaging tests to better determine if that suspicious feature might be breast cancer. These additional imaging tests include repeated mammograms, magnification mammograms and/or ultrasound. Depending on what is seen in these images, the radiologist will provide a diagnosis that the suspicion is probably cancer, probably benign, or that the suspicion is a "false alarm." If it is a false alarm, then the woman is sent home and she should come back after a year for another standard annual mammogram. If the diagnosis is that it is probably benign, then the woman should come back after 6 months so that the suspicion can be tested again. If the diagnosis is that it is probably cancer, the woman is recommended to have a biopsy so that the cancer can be confirmed. Both fortunately and unfortunately, 80% of the biopsies turn out to be "false alarms." Although confirming that a woman does not have cancer is always a very good thing, having put her through the anxiety, expense, and risk of a biopsy for what turned out to be nothing should be avoided. Therefore, it would be desirable to reduce the number of unnecessary biopsies that are performed.

Dedicated breast computed tomography (or breast CT), a new way of imaging the breast, has been introduced in the last few years. Breast CT is an x-ray exam that uses 3D imaging to show the breast in its real three dimensional shape. The investigators propose to use breast CT as a new, better tool for the radiologist to perform the diagnosis, and therefore hopefully result in fewer biopsies, which should decrease the "false alarms." Before breast CT can be used clinically as a diagnostic tool, extensive testing must be performed. In this first step, the investigators propose to acquire breast CT images of only 10 patients that have been recommended to have biopsies, to see if the radiologist would have arrived at a different diagnosis if he/she had based his/her decision on the breast CT images. Since this has never been attempted before, this is an initial small study to test the feasibility of this method.

DETAILED DESCRIPTION:
See Brief Summary

ELIGIBILITY:
Inclusion Criteria:

* All subjects will be women at least 35 years of age that have been found, after diagnostic workup, to have focal distributions of microcalcifications (BI-RADS 4 or 5) or focal soft tissue lesions (BI-RADS 4 or 5)

Exclusion Criteria:

* Subject does not meet any of the inclusion criteria
* Women with suspected or confirmed pregnancy
* Women who have had bilateral mastectomy
* Women who are very frail and unable to cooperate
* Women who are under 35 years of age
* Women who cannot give informed consent
* Male subjects
* Women with implants
* Subject has had breast augmentation, except for unilateral augmentation done for prior mastectomy
* Women recalled for bilateral workup
* Women with physical limitations such as, but not limited to: frozen shoulder, recent heart surgery, pace maker, neck problems, or any other condition that would prohibit them from lying face down

Min Age: 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Women having breast biopsy for either masses or calcifications
Sampling Method: Non-Probability Sample
Enrollment: 16 (Actual)
Dates: Start 2009-05; Primary Completion 2010-01 (Actual); Study Completion 2015-01 (Actual)

PRIMARY OUTCOMES:
Reduction in negative biopsies | After biopsy

CONTACTS AND LOCATIONS:
Overall Officials: Ioannis Sechopoulos, PhD, Principal Investigator — Emory University
Locations (1):
- Emory University Hospital Breast Imaging Center, Atlanta, Georgia, United States